CLINICAL TRIAL: NCT05891990
Title: Evaluation of Soft and Hard Tissue Changes After Immediate Implant Placement With Sticky Tooth Versus Autogenous Tooth Graft In Cases With Labial Plate Dehiscence: A 1-Year Randomized Clinical Trial
Brief Title: Immediate Implant Placement With Sticky Tooth Versus Autogenous Tooth Graft In Cases With Labial Plate Dehiscence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Halla Gamal Mohammed Esmail (Other)
Responsible Party: Sponsor-Investigator, Halla Gamal Mohammed Esmail, Dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023
Record Dates: First submitted 2023-05-27; First posted 2023-06-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Immediate Implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): sticky tooth preparation:
  * patient's venous blood will be collected using a 21 g needle with a butterfly handle.
  * The blood in the test tubes will be centrifuged at 700 rpm for 3 min for women and 4 min for men because of a different hematocrit.
  * The liquid PRF fraction will be collected using a sterile syringe. It gently will be mixed with the demineralized dentin granules and allowed for five-ten minutes for polymerization in order to produce a sticky tooth.
  Interventions: Procedure: immediate implant augmented with sticky tooth
- Control group (Active Comparator): Autogenous demineralized dentin graft preparation
  * Extracted teeth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries, or restorations (if present), using a high-speed fine finishing stone and saline irrigation.
  * The pulp will be removed, using a root canal instrument. Subsequently, the remaining dentin will be cut into pieces. These pieces of dentin will be ground using a bone mill to produce dentin particles.
  * The sorted particles will be immersed in 70% ethanol and 4% H2O2 in a sterile container to remove any soft tissue remnants, bacteria, and smear layer.
  * Tooth particles will be demineralized using 0.6N HCl for 30 minutes to expose the dentine organic matrix.
  * After demineralization, the materials will be washed with phosphate-buffered saline (PBS) and dried with sterile gauze.
  Interventions: Procedure: immediate implant augmented with autogenous tooth graft

INTERVENTIONS:
Procedure: immediate implant augmented with sticky tooth — * Topical anesthesia will be administered using an infiltration technique.
  * Atraumatic extraction will be done with the aid of periotome and Luxators.
  * The extraction socket will be debrided to remove any residual debris or granulation tissue.
  * Full-thickness midcrestal incision and vertical releasing incision on the distal side will be made, and a vertical releasing incision on the mesial side will be made if necessary. The extraction socket and the labial bone defect will be exposed by buccal and palatal flap reflection.
  * Implant insertion will be performed according to the manufacturer's instruction, and then the implant will be inserted 2mm apical to the alveolar bone crest with adequate primary stability.
  * The gap between the implant and the defect of the facial bone will be filled with the sticky tooth to reach enough buccal bone supported and then will be covered with absorbable barrier collagen membranes.
  * Finally, the flap will be repositioned and sutured.
  Arms: Intervention group
Procedure: immediate implant augmented with autogenous tooth graft — * Topical anesthesia will be administered using an infiltration technique.
  * Atraumatic extraction will be done with the aid of periotome and Luxators.
  * The extraction socket will be debrided to remove any residual debris or granulation tissue.
  * Full-thickness midcrestal incision and vertical releasing incision on the distal side will be made, and a vertical releasing incision on the mesial side will be made if necessary. The extraction socket and the labial bone defect will be exposed by buccal and palatal flap reflection.
  * Implant insertion will be performed according to the manufacturer's instruction, and then the implant will be inserted 2mm apical to the alveolar bone crest with adequate primary stability.
  * The gap between the implant and the defect of the facial bone will be filled with the autogenous demineralized dentin graft to reach enough buccal bone supported and then will be covered with collagen membranes.
  * Finally, the flap will be repositioned and sutured.
  Arms: Control group

SUMMARY:
Evaluation of Soft and Hard Tissue Changes After Immediate Implant Placement With Sticky Tooth Versus Autogenous Tooth Graft for management of Cases With Labial Plate Dehiscence

DETAILED DESCRIPTION:
In patients with labial plate dehiscence in the esthetic zone, there is no difference between the use of tooth-derived granules in combination with platelet-rich fibrin ("sticky tooth") and autogenous tooth graft in conjunction with immediate implant placement in enhancing the amount of bone labial to the implant

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable teeth in the esthetic zone with a defect of labial bone.

  * Teeth with no acute inflammation.
  * Patients are free from any systemic condition that may affect the healing.
  * Availability of bone apical and palatal to the socket to provide primary stability
  * Good oral health.
  * Willingness to sign the informed consent form.

Exclusion Criteria:

* Heavy smoker (> 10 cigarettes/day)
* Pregnant females
* Contraindication for Implant surgery.
* Patients with poor oral hygiene.
* Acute inflammation in the site of implantation and adjacent tissue.
* A history of radiotherapy in the head or neck region.
* Patients with systemic diseases like uncontrolled diabetes mellitus, coagulation disorders, alcohol or drug abuse not suitable for implantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic width of bone labial to the implant | 1 year
  Amount of bone labial to the implant will be measured perpendicular to the vertical line of the implant surface at the implant neck level or the top of the buccal bone (which is regarded as 0 mm), 3 mm and 6 mm apical to the implant neck Each measurement will be recorded at different times

SECONDARY OUTCOMES:
Radiographic horizontal bucco-palatal bone changes | 1 year
  The bucco-palatal width of the alveolar bone will be measured perpendicular to the long axis of the alveolar bone; the 3 measurements will be the coronal width (CW), middle width (MW), and apical width (AW). Each measurement will be recorded at different times
Radiographic vertical bone changes | 1 year
  Vertical bone height will be measured. Measurement will be taken at highest point of the remaining labial/buccal plate of bone using the implant neck as a reference point. Each measurement will be recorded at different times and the difference between pre and post-operative measurements will be determined as the gain in labial/buccal vertical bone dimension
Esthetic evaluation (The pink esthetic score) | 1 year
  The pink esthetic score will be calculated on the parameters defined by (Fürhauser et al. 2005). Clinical photographs will be taken to evaluate peri-implant soft tissue through evaluating seven variables compared to a natural reference tooth including: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value. The maximum achievable PES is 14.
Implant stability | 6 months
  Implant stability will be measured using Ostell which has a scale ranges from 1 to 100, the higher the ISQ the more stability
Gingival Thickness | 1 year
  Gingival thickness will be evaluated 2 mm below the gingival margin with a short needle for and silicon disk stop. The needle will be inserted perpendicular to the mucosal surface, through the soft tissues with light pressure until a hard surface was reached. The silicone disc stop was then mounted in close contact with the gingival tissue surface. The insertion depth was assessed with a digital caliper accurate to the nearest 0.1 mm
Width of the Keratinized Tissue | 1 year
  It will be evaluated from the gingival margin to the mucogingival junction (MGJ). The MGJ was assessed with roll technique
Midfacial recession | 1 year
  Corono-apical distance between the peri-implant soft tissue margin and the cemento-enamel junction (CEJ) of the homologous contralateral tooth
Post-Operative Pain | 7 days
  Pain will be assessed post-surgically using the Visual Analogue Scale (VAS) with numbers from 0 to 10 score zero represented no pain while score 10 represented the worst pain imaginable
Post-Operative patient's Satisfaction | 1 year
  Three Yes or No Questions will be asked to the patient about his overall satisfaction about the procedure
  /
Post-operative swelling | 7 days
  Swelling will be assessed post-surgically using the Verbal Rating Scale (VRS) (García et al. 2008):
  * Absent (no swelling),
  * Slight (intraoral swelling at the operated area),
  * Moderate (moderate intraoral swelling at the operated area) and
  * Intense (intensive extraoral swelling extending beyond the operated area)

IPD SHARING:
Plan to Share IPD: Undecided